CLINICAL TRIAL: NCT03213665
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of Tazemetostat in Patients With Tumors Harboring Alterations in EZH2 or Members of the SWI/SNF Complex
Brief Title: Tazemetostat in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With EZH2, SMARCB1, or SMARCA4 Gene Mutations (A Pediatric MATCH Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01245; NCI-2017-01245 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621C; APEC1621C (Other: Children's Oncology Group); APEC1621C (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Hodgkin Lymphoma; Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma; Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Low Grade Glioma; Recurrent Ependymoma; Recurrent Ewing Sarcoma; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Hodgkin Lymphoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Glioma; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Primary Central Nervous System Neoplasm; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Refractory Hodgkin Lymphoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Rhabdoid Tumor; Refractory Soft Tissue Sarcoma; Rhabdoid Tumor; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Wilms Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral; Ependymoma; Sarcoma, Ewing; Glioma; Hepatoblastoma; Hodgkin Disease; Histiocytosis, Langerhans-Cell; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Central Nervous System Neoplasms; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Wilms Tumor | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tazemetostat) (Experimental): Patients receive tazemetostat PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Given PO
  Other Names: E 7438; E-7438; E7438; EPZ 6438; EPZ-6438; EPZ6438

SUMMARY:
This phase II Pediatric MATCH trial studies how well tazemetostat works in treating patients with brain tumors, solid tumors, non-Hodgkin lymphoma, or histiocytic disorders that have come back (relapsed) or do not respond to treatment (refractory) and have EZH2, SMARCB1, or SMARCA4 gene mutations. Tazemetostat may stop the growth of tumor cells by blocking EZH2 and its relation to some of the pathways needed for cell proliferation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with tazemetostat with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphoma or histiocytic disorders that harbor gain of function mutations in EZH2, or loss of function mutations in the SWI/SNF complex subunits SMARCB1 or SMARCA4 at a dose of 520 mg/m^2/dose twice daily for patients without any CNS involvement or 1200 mg/m^2/dose orally twice daily for patients with CNS involvement.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival in pediatric patients treated with tazemetostat that harbor gain of function mutations in EZH2, or loss of function mutations in the SWI/SNF complex subunits SMARCB1 or SMARCA4.

II. To obtain information about the tolerability of tazemetostat in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate other biomarkers as predictors of response to tazemetostat and specifically, whether tumors that harbor different missense mutations or fusions will demonstrate differential response to tazemetostat treatment.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive tazemetostat orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621C based on the presence of an actionable mutation
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have MIBG+ evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) and visible on more than one slice; Note: The following do not qualify as measurable disease:

  * Malignant fluid collections (e.g., ascites, pleural effusions)
  * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
  * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
  * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
  * Previously radiated lesions that have not demonstrated clear progression post radiation
  * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation; Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have had prior exposure to tazemetostat or other inhibitor(s) of EZH2
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: male: 0.6 mg/dL; female: 0.6 mg/dL
  * Age 2 to < 6 years: male: 0.8 mg/dL; female: 0.8 mg/dL
  * Age 6 to < 10 years: male: 1 mg/dL; female: 1 mg/dL
  * Age 10 to < 13 years: male: 1.2 mg/dL; female: 1.2 mg/dL
  * Age 13 to < 16 years: male: 1.5 mg/dL; female: 1.4 mg/dL
  * Age >= 16 years: male: 1.7 mg/dL; female: 1.4 mg/dL
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Corrected QT (QTc) interval =< 480 milliseconds
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [V] 4.0) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible
* International normalized ratio (INR) =< 1.5
* For subjects with CNS involvement (primary tumor or metastatic disease): Subjects must not have any active bleeding, or new intratumoral hemorrhage of more than punctate size on screening MRI or known bleeding diathesis or treatment with anti-platelet or anti-thrombotic agents
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study because there is currently no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study treatment; female subjects of childbearing potential should agree to remain abstinent or use adequate contraceptive methods for 30 days after the last dose of tazemetostat; male subjects should agree to remain abstinent or use adequate contraceptive methods, and agree to refrain from donating sperm, and for 90 days after the last dose of tazemetostat
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are strong inducers or strong inhibitors of CYP3A4 are not eligible; strong inducers or inhibitors of CYP3A4 are prohibited from 14 days prior to the first dose of tazemetostat to the end of the study; Note: Dexamethasone for CNS tumors or metastases, on a stable dose, is allowed
* Patients who have an uncontrolled infection are not eligible
* On complete blood count (CBC) differential, patients must not have any significant morphologic abnormalities concerning for myeloproliferative neoplasm (MPN)/myelodysplastic syndrome (MDS) or T- acute lymphoblastic leukemia (ALL)
* Patients must not have thrombocytopenia, neutropenia, or anemia of grade >= 3 (per CTCAE 5.0 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)
* Patients with a history of prior history of T-lymphoblastic lymphoma (LBL)/T-ALL
* Patients with any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).
* Patients who have received prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N Chi, Principal Investigator — Children's Oncology Group
Locations (117):
- United States (115):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Tazemetostat)
Started | 20
Completed | 1
Not Completed | 19
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 13

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tazemetostat)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR will be defined as complete response + partial response and assessed by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.
Time Frame: From enrollment to the end of treatment, up to 2 years
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Tazemetostat)
Number analyzed (Participants) | 20
Percentage of participants | 5 [1 to 20]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free survival will be defined as time from the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause. PFS along with the confidence intervals will be estimated using the Kaplan-Meier method.
Time Frame: From start of subprotocol treatment to time of progression or death, whichever occurs first, assessed for up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tazemetostat)
Number analyzed (Participants) | 20
percentage of participants | 35 [15.7 to 55.2]

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or 4 Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Any eligible patient who receives at least one dose of protocol therapy will be considered in the evaluation of toxicity. A patient will be counted only once for a given toxicity for the worst grade of that toxicity reported for that patient.
Time Frame: From initiation of treatment to disease progression, disease recurrence, or death from any cause assessed up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tazemetostat)
Number analyzed (Participants) | 20
percentage of participants | 90 [68.3 to 98.8]

4. Other Pre Specified Outcome: Biomarker Predictors of Response to Tazemetostat
Description: Will evaluate other biomarkers as predictors of response to tazemetostat and specifically, whether tumors that harbor different missense mutations or fusions will demonstrate differential response to tazemetostat treatment. Will be performed and will be summarized with simple summary statistics and will be descriptive in nature.
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Tumor Genomics
Description: To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid. Will be performed and will be summarized with simple summary statistics and will be descriptive in nature.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to 30 days after the end of treatment, up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Tazemetostat)
All-Cause Mortality (participants affected / at risk) | 7/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tazemetostat) (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 6
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hydrocephalus (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Muscle weakness right-sided (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tazemetostat) (N=20)
Anemia (Blood and lymphatic system disorders) | 9
Eosinophilia (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Cushingoid (Endocrine disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Edema face (General disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 10
Fever (General disorders) | 5
Gait disturbance (General disorders) | 1
Generalized edema (General disorders) | 2
Hypothermia (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 2
Fibrinogen decreased (Investigations) | 1
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
Weight gain (Investigations) | 2
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Oculomotor nerve disorder (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT03213665/Prot_SAP_000.pdf